CLINICAL TRIAL: NCT04411888
Title: Observation Study of Clinical Manifestation and Outcome in Chinese Pulmonary Embolism
Brief Title: Pulmonary Embolism Prognosis Model
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH--Pulmonary embolism
Record Dates: First submitted 2020-05-24; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observation — observation

SUMMARY:
The purpose of this study is to analyze the clinical manifestations, imaging features, and prognosis-related factors of pulmonary embolism, and to explore the prognosis risk assessment model for Chinese patients

DETAILED DESCRIPTION:
Patients with pulmonary embolism and aged 18 years or older were enrolled in this study.Patient demographic characteristics((age, sex, department, diagnosis, ), basic vital signs, symptoms at their admissions (hemoptysis, dyspnea, chest pain, syncope), laboratory examinations (blood lab routines, blood gas, liver and kidney function, myocardial marker), and imaging examinations (vascular ultrasonography, computed tomographic angiography, echocardiography, chest CT, CTPA, pulmonary perfusion imaging, pulmonary angiography, PET/CT) were collected by reviewing the cases. The prognostic information was collected by telephone follow-up. The follow-up end point was June 2024.

ELIGIBILITY:
Inclusion Criteria:

Aged 18 years or older. Discharged with the diagnosis of PE from Peking Union Medical College Hospital.

Exclusion Criteria:

Diagnosed PE by other health care facility or transferred from other health care facility .

Without important follow-up data.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients diagnosed as pulmonary embolism who meet the inclusion criteria above.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient survival time | Through study completion, an average of 4 year
  Patient survival time after diagnosed as pulmonary embolism

CONTACTS AND LOCATIONS:
Overall Officials: Juhong Shi, M.D, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China